CLINICAL TRIAL: NCT02846025
Title: Profile Of Methylation and Gene Expression Of Gene ADRB3 And Effects Of Ingestion Of Folate, Hazelnuts And Diets Oil Capsule Antioxidants In Case Inflammatory
Brief Title: Profile Of Methylation and Gene Expression Of Gene ADRB3 And Effects Of Folate Intake
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Raquel Patricia Ataide Lima, Master, Federal University of Paraíba
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: UFPBNUTRI
Record Dates: First submitted 2016-07-15; First posted 2016-07-27 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Folic Acid; Antioxidants

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Folate (Other): diet rich in folate
  Interventions: Dietary Supplement: Folate and capsule of oil hazel; Dietary Supplement: Folate and placebo
- placebo (Other): placebo
  Interventions: Dietary Supplement: Folate and placebo; Dietary Supplement: antioxidant and placebo
- diet antioxidant (Other): diet antioxidant
  Interventions: Dietary Supplement: antioxidant and placebo
- Hazelnut Oil (Other): hazelnut oil capsule
  Interventions: Dietary Supplement: Folate and capsule of oil hazel

INTERVENTIONS:
Dietary Supplement: Folate and capsule of oil hazel — rich diet aministracao folate and capsule of oil hazel
  Arms: Folate; Hazelnut Oil
Dietary Supplement: Folate and placebo — rich diet aministracao folate and placebo
  Arms: Folate; placebo
Dietary Supplement: antioxidant and placebo — antioxidant diet (90μg folate) and placebo capsule
  Arms: diet antioxidant; placebo

SUMMARY:
ABSTRACT

Epigenetic mechanisms may be involved in the regulation of lipid metabolism and inflammatory markers may therefore contribute to the cardiovascular risk profile, as well as environmental factors have a significant impact on the epigenetic program of gene expression. Methyl groups are usually added or removed as needed and can be influenced by diet soon, dietary factors have been linked to the change of DNA methylation, resulting in changes in gene expression. Research on the prevalence of gene methylation levels on the impact of nutrient intake, as well as the inflammatory condition and the results of dietary interventions for the genes, it is a sparse area in studies and, therefore, expanding of the knowledge. Thus, understanding the effects of a diet rich in antioxidants and hazelnut oil, in inflammation and DNA methylation profile is important because chronic diseases with cardiovascular disease can begin with the consumption of modified lipids and can research this stage provide important dietary allowances for the development of this disease prevention strategies even in adulthood. This PhD project is linked to a larger project entitled "II Diagnosis Cycle and Intervention Food Situation, Nutrition and Noncommunicable Diseases Prevalent over the City Population of João Pessoa / PB" (II DISANDNT / PB) and have two methodological designs: the first one is the composition of a representative sample of adults in the city of João Pessoa, from II DISANDNT / JP, population-based study and cross-sectional. The second methodological design was developed with a subsample of the above population, selected from criteria being the type and interventional clinical trial. This model will have to evaluate the effect of a diet rich in antioxidant and hazelnut oil, in inflammation and gene expression.

DETAILED DESCRIPTION:
This thesis is linked to a population-based survey entitled "Diagnosis II Cycle and Intervention Food Situation, Nutrition and Noncommunicable Diseases Prevalent over the city of João Pessoa Population / PB" (II DISANDNT / PB).

For realization of this thesis, a first population-based study, representative of adults in the east areas and west of the city of João Pessoa, there was the calculation of a representative sample for the age group of adults, using information provided by the city, as map the municipality, the number of blocks per district and the Brazilian Institute of Geography and Statistics.

Home visits and implementation of the survey questionnaires were carried out by teams of undergraduate researchers from the Nutrition courses, masters and doctoral students of the Post Graduate Program in Nutrition Sciences (PPGCN) UFPB duly previously trained at the beginning of data collection after the pilot study and following.

The trained teams, after recognizing the drawn court, were instructed to select all households in the court. The blocks that did not have homes, the homes in which those responsible have not accepted to participate and the amount of individuals who refused to participate in randomly selected households were computed and resorteadas randomly thereafter to minimize losses.

In each residence drawn all individuals, adults aged between 20-59 years were invited to participate in the research through application of socioeconomic and demographic characteristics questionnaires, epidemiological characterization, nutritional assessment and food intake, biochemical evaluation and brands epigenetic.

ELIGIBILITY:
Inclusion Criteria:

* Individuals adults, aged 20 and 59 years;
* Being female;
* Individuals who have hypermethylation in ADRB3 gene;
* cognitive state preserved.

Exclusion Criteria:

* Individuals drinkers or smokers;

  * Take medications known to interfere with the metabolism of folic acid (the last 3 months);
  * Individuals who make use of fish oil supplement or other fatty acids;
  * Pregnant or planning to become pregnant during the study period.

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in value of the weight (kg) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria José Carvalho Costa, Doctor, Study Director — UFPB

IPD SHARING:
Plan to Share IPD: Yes
The data of the participants are in the excel database

REFERENCES:
- [Derived] Lima RPA, do Nascimento RAF, Luna RCP, Persuhn DC, da Silva AS, da Conceicao Rodrigues Goncalves M, de Almeida ATC, de Moraes RM, Junior EV, Fouilloux-Meugnier E, Vidal H, Pirola L, Magnani M, de Oliveira NFP, Prada PO, de Carvalho Costa MJ. Effect of a diet containing folate and hazelnut oil capsule on the methylation level of the ADRB3 gene, lipid profile and oxidative stress in overweight or obese women. Clin Epigenetics. 2017 Oct 13;9:110. doi: 10.1186/s13148-017-0407-6. eCollection 2017. PMID 29046732